CLINICAL TRIAL: NCT00579111
Title: Reduced-Intensity Preparative Regiment With Fludarabine, Busulfan, And Alemtuzumab (Campath 1H) Followed By Allogeneic Hematopoietic Stem Cell Transplant For Malignant And Non-Malignant Hematological Diseases
Brief Title: Reduced Intensity Preparative Regimen Followed by Stem Cell Transplant (FAB)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Rammurti Kamble, Associate Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19386; FAB; NCT00625144 (obsolete NCT alias)
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2012-08-09 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-03

CONDITIONS: Myelodysplastic and Myeloproliferative Disorders; Acute Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Chronic Myelogenous Leukemia; Multiple Myeloma; Plasma Cell Dyscrasia; Lymphoproliferative Disorders; Hematologic Diseases
Keywords: Myelodysplastic and Myeloproliferative Disorders; Acute Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Chronic Myelogenous Leukemia; Multiple Myeloma; Plasma Cell dyscrasia; Lymphoproliferative disorders; Hematologic Diseases; Fludarabine; Busulfan; Campath; Alemtuzumab; allogeneic stem cell transplant
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Multiple Myeloma; Paraproteinemias; Lymphoproliferative Disorders; Hematologic Diseases | interventions — Alemtuzumab; Busulfan; fludarabine; Stem Cell Transplantation; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HLA-identical sibling transplant (Experimental): Recipients of HLA identical sibling stem cell transplants
  Interventions: Drug: Campath; Drug: Busulfan; Drug: Fludarabine; Procedure: Hematopoietic stem cell infusion; Drug: FK-506
- Unrelated Matched or Single Antigen Mismatched transplant (Experimental): Recipients of unrelated matched or single antigen mismatched donor stem cell transplant or single antigen mismatched family donor stem cell transplants
  Interventions: Drug: Campath; Drug: Busulfan; Drug: Fludarabine; Procedure: Hematopoietic stem cell infusion; Drug: FK-506

INTERVENTIONS:
Drug: Campath — 10 mg/day IV daily for 3 days on days -6 to D-4. Campath may be omitted from the conditioning regimen for patients with malignant diseases and matched related donor transplants
  Other Names: Alemtuzumab
Drug: Busulfan — 3.2 mg/kg/day IV daily for 2 days, infused over 3 hours, on Day -5 and Day -4
Drug: Fludarabine — 30mg/m2/day IV daily for 4 days on Day -5 to D -2
Procedure: Hematopoietic stem cell infusion — Peripheral blood stem cells when possible. Bone marrow cells will be used if peripheral blood cells are insufficient or unavailable.
Drug: FK-506 — FK-506 at a dose of 0.03 mg/kd/day will be administered via continuous infusion over 24 hours from 4pm on Day -2 until engraftment or when the patient is able to take PO, then 0.03 mg/kg PO every 12 hours.
  Other Names: Tacrolimus

SUMMARY:
Blood disorders such as leukemia or lymphoma or hemoglobinopathies can benefit from receiving an allogeneic (meaning that the cells are from a donor) stem cell transplant. Stem cells are created in the bone marrow. They grow into different types of blood cells that the body needs, including red blood cells, white blood cells, and platelets. In a transplant, the body's stem cells would be killed and then replaced by stem cells from the donor. Usually, patients are given very high doses of chemotherapy (drugs which kill cancer cells) prior to receiving a stem cell transplant. However, patients that are older, have received several prior treatments, or have other organ diseases are at a high risk of getting life-threatening treatment-related side effects from high doses of chemotherapy. Over the past several years, some doctors have begun to use lower doses of chemotherapy for preparing patients for a stem cell transplant.

A condition that can occur after a stem cell transplant from a donor is Graft Versus Host Disease (GVHD). It is a rare but serious disorder that can strike persons whose immune system is suppressed and have received either a blood transfusion or a bone marrow transplant. Symptoms may include skin rash, intestinal problems similar to inflammation of the bowel and liver dysfunction.

This research study uses a combination of lower-dose chemotherapy agents that is slightly different from those that have been used before.

The medicines that will be used in this study are Fludarabine, Busulfan, both chemotherapy medicines, and Campath. Campath is a monoclonal antibody (a type of substance produced in the laboratory that binds to cancer cells). It helps the immune system see the cancer cell as something that needs to be destroyed.

This research study will help us learn if using Fludarabine, Busulfan and Campath prior to an allogeneic stem cell transplant can provide treatment for blood disorders while decreasing the incidence of side effects.

DETAILED DESCRIPTION:
Allogeneic stem cell transplantation with high-dose chemotherapy affords a better chance of cure of malignant and non-malignant hematological diseases compared to autologous transplantation, because of the lack of stem cell contamination and the immune mediated graft vs. leukemia effect. Unfortunately, high-dose chemotherapy and allogeneic stem cell transplantation has a substantial treatment related mortality, that is particularly high in older patients (greater than 50 yrs of age), or in those with co-morbidities such as congestive heart disease and pulmonary disease. Patients who have pre-existing infections or who have had multiple relapses with prior chemotherapy are also at high risk. In all these groups, treatment related mortality may exceed 50%, making them ineligible for high-dose chemotherapy and allogeneic stem cell transplantation.

Recently interest has increased in using less toxic chemotherapy protocols that are termed submyeloablative. The intent is to allow partial engraftment of a donor immune and hemopoietic systems with subsequent progressive replacement of the host's own hemopoiesis and immunity. As the donor immune system becomes established, patients may develop full donor chimerism, without passing through the period of prolonged aplasia associated with conventional conditioning regimens, and with less of the associated toxicity. Preliminary results in high-risk patients have shown treatment related mortality (TRM) of 15-20%, versus 50% expected, with an overall survival rate of 70-80% at 1-2 years post transplant.

As might be anticipated, the major problem with sub-ablative conditioning is that the graft failure rate is increased, with published figures of 5-30% versus 1-5% predicted in fully ablated patients. The incorporation of lymphodepleting antibodies in the preliminary conditioning regimen may allow these rejection rates to be diminished. Moreover, a highly efficient lymphodepleting MAb or MAb combination might be successfully substituted in part or in whole for cytotoxic and immunosuppressive drugs, further increasing the safety and efficacy of the subablative approach to stem cell transplantation. Our own data using the crude polyclonal mixture of antibodies in ATG as a component of pre-transplant conditioning revealed an improvement in engraftment during matched unrelated donor transplantation.The lymphodepleting monoclonal antibody Campath IH has many of the properties desired for this application, and we propose to incorporate it in our conditioning regimen. Since CAMPATH1H persists after infusion, we would expect it to have additional anti-GvHD effector function, further reducing treatment related mortality (TRM).

The following preparative regimen will be delivered to all patients:

1. Busulfan 3.2 mg/kg/day IV daily for 2 days, infused over 3 hours, on Day -5 and Day -4
2. Fludarabine 30mg/m2/day IV daily for 4 days on Day -5 to D -2
3. Campath 10 mg/day IV daily for 3 days on days -6 to D-4.

Because CAMPATH-1H infusions will provide a persisting level of antibody over the transplant period, it will contribute to anti-GvHD activity. Additional Graft vs. host disease prophylaxis will consist of FK506 administered from Day-2.

The stem cells will be infused on day 0.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of myelodysplastic and myeloproliferative disorders, acute myelogenous leukemia, acute lymphoblastic leukemia, chronic myelogenous leukemia, multiple myeloma, plasma cell dyscrasia, lymphoproliferative disorders (non-Hodgkin lymphoma, hairy cell leukemia, chronic lymphocytic leukemia, and Hodgkin's disease) and non malignant hematologic diseases considered treatable with an allogeneic transplant including but not limited to bone marrow failure syndrome, hemoglobinopathy and severe immunodeficiency states.
2. Performance status 0-2 on Zubrod scale
3. Ejection fraction > 30%
4. AST/ALT and bilirubin not > 4 times normal
5. FEV1 greater than 1.0 and diffusion capacity > 40%
6. Age birth to 70 years of age
7. Conditions that increase treatment related mortality (need more than one to be eligible):

   * Age > 35 years
   * EF of less than 45%
   * DLCO less than 50% or FEV1 50-75% of predicted value
   * Diabetes mellitus
   * Renal insufficiency, defined by increase in serum creatinine level of 1.5 times ULN or decrease in GFR by 25%
   * Prior recent history of systemic fungal infection
   * 3rd or greater remission of AML or ALL
   * More than 1 year of diagnosis (CML or myeloma patients only)
   * Multiple types of treatment regimens (equal to or more than 3)
   * Prior autologous or allogeneic stem cell transplantation
   * Significant Grade III or IV neurologic or hepatic toxicity as defined by NCI CTC toxicity from previous treatment
   * No matched sibling donor
8. Available healthy donor without any contraindications for donation

   * 5/6 or 6/6 related
   * 5/6 or 6/6 unrelated (molecular typing for DRB1)
9. Patient and/or responsible person able to understand and sign consent
10. For women of childbearing potential, negative pregnancy test

Exclusion Criteria:

1. Pregnant and lactating women or women unwilling to use contraception.
2. HIV positive patient.
3. Uncontrolled intercurrent infection.
4. Refractory AML or ALL.
5. Untreated blast crisis for CML.
6. Uncontrolled high-grade lymphoproliferative disease/lymphoma.
7. Unstable angina and uncompensated congestive heart failure (Zubrod of 3 or greater).
8. Severe chronic pulmonary disease requiring oxygen (Zubrod of 3 or greater).
9. Hemodialysis dependent.
10. Active Hepatitis or cirrhosis with total bilirubin, SGOT, and SGPT greater than 3 x normal.
11. Serum creatinine >2x ULN.
12. Unstable cerebral vascular disease and recent hemorrhagic stroke (less than 6 months).
13. Active CNS disease from hematological disorder.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-06; Primary Completion 2009-02 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rammurti T Kamble, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HLA-identical Sibling Transplant | Unrelated Matched or Single Antigen Mismatched Transplant
Started | 3 | 1
Completed | 1 | 0
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HLA-identical Sibling Transplant | Unrelated Matched or Single Antigen Mismatched Transplant | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Customized [Number; unit: participants]
  Between 50 and 65 years | 3 | 0 | 3
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Successful Donor Engraftment
Description: Each patient will be classified as a success or failure. A success will be defined as engraftment of at least 35% of cells 100 days after transplant.
Time Frame: 100 days
Measure: Number; unit: participants
Arm/Group | HLA-identical Sibling Transplant | Unrelated Matched or Single Antigen Mismatched Transplant
Number analyzed (Participants) | 3 | 1
participants | 2 | 1

2. Secondary Outcome: Number of Patients With Treatment Related Grade III or IV Non-hematological Toxicity
Time Frame: 100 days
Measure: Number; unit: participants
Arm/Group | HLA-identical Sibling Transplant | Unrelated Matched or Single Antigen Mismatched Transplant
Number analyzed (Participants) | 3 | 1
participants | 1 | 0

ADVERSE EVENTS:
Arm/Group | HLA-identical Sibling Transplant | Unrelated Matched or Single Antigen Mismatched Transplant
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/1
Other Adverse Events (participants affected / at risk) | 0/3 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HLA-identical Sibling Transplant (N=3) | Unrelated Matched or Single Antigen Mismatched Transplant (N=1)
Blood/Bone Marrow - Other: Engraftment Failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e (Infections and infestations) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes